CLINICAL TRIAL: NCT01030523
Title: Study on ASTRA TECH Implant System, Short Implants (OsseoSpeed™) Compared to Standard Length Implants (OsseoSpeed™) in Combination With Bone Grafting
Brief Title: Short Implants - An Alternative to Bone Grafting?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-SHO-0002
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially | interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Short Implants (Experimental): ASTRA TECH Implant System, OsseoSpeed™ 4.0 S (length: 6 mm)
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™ 4.0 S (length: 6 mm)
- Long Implants in combination with bone grafting (Active Comparator): ASTRA TECH Implants System, OsseoSpeed™ implants (lengths: 11, 13, 15 mm) in combination with bone grafting
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™ implants (lengths: 11, 13, 15 mm) in combination with bone grafting

INTERVENTIONS:
Device: ASTRA TECH Implant System, OsseoSpeed™ 4.0 S (length: 6 mm) — ASTRA TECH Implant System, OsseoSpeed™ 4.0 S (length: 6 mm)
  Arms: Short Implants
Device: ASTRA TECH Implant System, OsseoSpeed™ implants (lengths: 11, 13, 15 mm) in combination with bone grafting — ASTRA TECH Implant System, OsseoSpeed™ implants (lengths: 11, 13, 15 mm) in combination with bone grafting
  Arms: Long Implants in combination with bone grafting

SUMMARY:
The study, with the ASTRA TECH Implant System, is comparing short implants (OsseoSpeed™) to standard length implants (OsseoSpeed™) in combination with bone grafting. The hypothesis is that the use of short implants in posterior maxilla with inadequate bone is as safe and predictable as placing standard length implants in combination with bone augmentation.

DETAILED DESCRIPTION:
This study was designed as an open, prospective, randomized, controlled, multicenter, 5-year follow-up investigation evaluating the outcome of treatment with the OsseoSpeed™ implant 6 mm placed in the posterior maxilla compared to treatment with OsseoSpeed™ implant 11, 13 or 15 mm placed after bone grafting. The study was during the conduct of the study amended to include a 10-year extension cohort.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Aged 20-75 years at enrolment
* History of edentulism in the study area of at least four months
* In need for 1-4 implants in either side of the posterior maxilla (premolar and molar region)
* Neighboring tooth/teeth to the planned implant/s must have natural root(s) or implant supported restoration, with absence of pathology or excessive bone loss, as judged by the investigator
* Presence of natural tooth/teeth, partial prosthesis and/or implants in the opposite jaw in contact with the planned crown/s
* Deemed by the investigator to have a bone height between 5 and 7 mm and a bone width of a minimum of 6 mm
* Deemed by the investigator as likely to present an initially stable implant situation

Exclusion Criteria:

* Unlikely to be able to comply with study procedures, as judged by the investigator
* Earlier bone graft procedures in the study area
* Uncontrolled pathologic processes in the oral cavity
* Known or suspected current malignancy
* History of radiation therapy in the head and neck region
* History of chemotherapy within 5 years prior to surgery
* Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration
* Uncontrolled diabetes mellitus
* Corticosteroids, iv bisphosphonates or any other medication that could influence post-operative healing and/or osseointegration
* Smoking more than 10 cigarettes/day
* Bruxism
* Present alcohol and/or drug abuse
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
* Previous enrolment in the present study
* Simultaneous participation in another clinical study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hämmerle, Prof. Dr., Principal Investigator — Zentrum für Zahn-, Mund- und Kieferheilkunde der Universität Zürich
Locations (5):
- Department of Oral Rehabilitation, Skeletal Development and Biomaterials, University of Connecticut, School of Dental Medicine, Farmington, Connecticut, United States
- Ärztegesellschaft für Zahn- Mund- und Kieferheilkunde, Akademie für Orale Implantologie: Fürhauser, Haas, Mailath-Pokorny & Watzek OG, Vienna, Austria
- Aesthetic Dent, Szczecin, Poland
- Facultad de Medicina y Odontologia, Universidade de Santiago de Compostela, Santiago de Compostela, Spain
- Zentrum für Zahn-, Mund- und Kieferheilkunde der Universität Zürich, Zurich, Switzerland

REFERENCES:
- [Result] Thoma DS, Haas R, Tutak M, Garcia A, Schincaglia GP, Hammerle CH. Randomized controlled multicentre study comparing short dental implants (6 mm) versus longer dental implants (11-15 mm) in combination with sinus floor elevation procedures. Part 1: demographics and patient-reported outcomes at 1 year of loading. J Clin Periodontol. 2015 Jan;42(1):72-80. doi: 10.1111/jcpe.12323. Epub 2014 Dec 26. PMID 25418606
- [Result] Schincaglia GP, Thoma DS, Haas R, Tutak M, Garcia A, Taylor TD, Hammerle CH. Randomized controlled multicenter study comparing short dental implants (6 mm) versus longer dental implants (11-15 mm) in combination with sinus floor elevation procedures. Part 2: clinical and radiographic outcomes at 1 year of loading. J Clin Periodontol. 2015 Nov;42(11):1042-51. doi: 10.1111/jcpe.12465. Epub 2015 Nov 27. PMID 26425812
- [Result] Pohl V, Thoma DS, Sporniak-Tutak K, Garcia-Garcia A, Taylor TD, Haas R, Hammerle CH. Short dental implants (6 mm) versus long dental implants (11-15 mm) in combination with sinus floor elevation procedures: 3-year results from a multicentre, randomized, controlled clinical trial. J Clin Periodontol. 2017 Apr;44(4):438-445. doi: 10.1111/jcpe.12694. Epub 2017 Mar 6. PMID 28081288
- [Result] Thoma DS, Haas R, Sporniak-Tutak K, Garcia A, Taylor TD, Hammerle CHF. Randomized controlled multicentre study comparing short dental implants (6 mm) versus longer dental implants (11-15 mm) in combination with sinus floor elevation procedures: 5-Year data. J Clin Periodontol. 2018 Dec;45(12):1465-1474. doi: 10.1111/jcpe.13025. Epub 2018 Nov 25. PMID 30341961
- [Derived] Thoma DS, Haas R, Sporniak-Tutak K, Garcia A, Taylor TD, Tutak M, Pohl V, Hammerle CHF. Randomized controlled multi-centre study comparing shorter dental implants (6 mm) to longer dental implants (11-15 mm) in combination with sinus floor elevation procedures: 10-year data. J Clin Periodontol. 2024 Apr;51(4):499-509. doi: 10.1111/jcpe.13954. Epub 2024 Jan 31. PMID 38296249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was amended to include a 10-year follow-up cohort where all subjects enrolled into the initial 5-year study were invited. In total 77 out of the initial 101 subjects consented and were enrolled into the 10-years extension cohort.
Units Other Than Participants: Implants
Period: Initial Study (5 Years)
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Started | 50; 67 Implants | 51; 70 Implants
Completed | 44; 60 Implants | 46; 64 Implants
Not Completed | 6; 7 Implants | 5; 6 Implants
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 4 | 5
Not completed — Implant failure | 1 | 0
Period: Follow-up Extension (10 Years)
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Started | 36; 48 Implants | 41; 57 Implants
Completed | 29; 39 Implants | 32; 47 Implants
Not Completed | 7; 9 Implants | 9; 10 Implants
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consists of all subjects enrolled into the study, n= 101.
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (12.88) | 50.5 (14.05) | 50.4 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 21 | 28 | 49

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival Rate
Description: Any implant that is removed after implant placement will be considered a failure, whatever the reason for removal. Implant survival will be evaluated clinically and radiographically by counting the number of remaining implants. Implant survival rate will be calculated by dividing the number of non-failures by the number of installed implant.
Time Frame: 5 years after permanent restoration
Population: Outcome measure only applicable for the initial study (5 years) cohort.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 50 | 51
Number analyzed (Implants) | 67 | 70
Implants | 66 | 70

2. Secondary Outcome: Average Marginal Bone Level (MBL) Change From Permanent Restoration on Implant Level
Description: Marginal bone level will be determined from radiographs and expressed as the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal bone level expressed in millimetres at the 5 year follow-up visit will be compared to values obtained at delivery of permanent restoration. Positive value denotes gain of bone. Negative value denotes loss of bone.
Time Frame: Time of permanent restoration and 5 years after permanent restoration
Population: Initial study (5 years) cohort. At visit 10 (5-year follow-up visit) 44 subjects remained in the short implants group, and 46 subjects remained in the long implants group. 10 subjects within the short implants group had missing or unreadable radiographs and could thus not be included in the analysis. The corresponding number for long implants group was 9 subjects with missing and unreadable radiographs.
Measure: Mean (Standard Deviation); unit: Millimetre
Units Other Than Participants: Implants
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 34 | 37
Number analyzed (Implants) | 44 | 49
Millimetre | -0.12 (0.535) | -0.18 (0.959)

3. Secondary Outcome: Average Marginal Bone Level (MBL) Change From Permanent Restoration on Implant Level
Description: Marginal bone level will be determined from radiographs and expressed as the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal bone level expressed in millimetres at the 10 year follow-up visit will be compared to values obtained for the 10-years cohort at delivery of permanent restoration. Positive value denotes gain of bone. Negative value denotes loss of bone.
Time Frame: Time of permanent restoration and 10 years after permanent restoration
Population: Follow-up Extension (10 years) cohort. At visit 15 (10-year follow-up visit) 29 subjects remained in the short implants group, and 32 subjects remained in the long implants group. 7 subjects within the short implants group had missing or unreadable radiographs and could thus not be included in the analysis. The corresponding number for long implants group was 9 subjects with missing and unreadable radiographs.
Measure: Mean (Standard Deviation); unit: Millimetre
Units Other Than Participants: implants
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 22 | 23
Number analyzed (implants) | 28 | 31
Millimetre | -0.12 (0.68) | -0.24 (0.82)

4. Secondary Outcome: Condition of Periimplant Mucosa Measured Through Bleeding on Probing (BoP)
Description: Bleeding on Probing will be evaluated at four aspects per implant, i.e. mesially, distally, buccally and palatinally by using a periodontal probe. BoP will be recorded as presence or absence (Yes or No) of bleeding when probing to the bottom of the pocket. The proportion of surfaces that show presence of bleeding will be calculated and presented on a subject level.
Time Frame: 5 years after permanent restoration
Population: Initial study (5 years) cohort. At visit 10 (5-year follow-up visit) 44 subjects remained in the short implants group, and 46 subjects remained in the long implants group. All subjects were included in the Intention-To-Treat population and were included in the analysis of BoP.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 44 | 46
Participants | 18 | 23

5. Secondary Outcome: Condition of Periimplant Mucosa Measured Through Bleeding on Probing (BoP)
Description: Bleeding on Probing will be evaluated at four aspects per implant, i.e. mesially, distally, buccally and palatinally by using a periodontal probe. BoP will be recorded as presence or absence (Yes or No) of bleeding when probing to the bottom of the pocket. The proportion of surfaces that show presence of bleeding will be calculated and presented on a subject level for the 10-years extension cohort.
Time Frame: 10 years after permanent restoration
Population: Follow-up Extension (10 years) cohort. At visit 15 (10-years follow-up visit) 29 subjects remained in the short implants group, and 32 subjects remained in the long implants group. All subjects were included in the ITT population and were included in the analysis of BoP.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 29 | 32
Participants | 16 | 23

6. Secondary Outcome: Condition of Periimplant Mucosa Measure by Average Change in Probing Pocket Depth (PPD) From Permanent Restoration
Description: PPD will be measured as the distance from the mucosal margin to the bottom of the probeable pocket in mm. A mean value will be calculated for each implant as well as for each subject. PPD changes in millimetres at the 5 year follow-up visit will be compared to values obtained at delivery of permanent restoration. Negative value denotes deeper pocket depth.
Time Frame: Time of permanent restoration and 5 years after permanent restoration
Population: Initial study (5 years) cohort. At visit 10 (5-year follow-up visit) 44 subjects remained in the short implants group, and 46 subjects remained in the long implants group. One subject in the short implants group did not have baseline PPD and was not included in the PPD analysis.
Measure: Mean (Standard Deviation); unit: Millimetre
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 43 | 46
Millimetre | -0.26 (0.91) | -0.43 (1.02)

7. Secondary Outcome: Condition of Periimplant Mucosa Measure by Average Change in Probing Pocket Depth (PPD) From Permanent Restoration
Description: PPD will be measured as the distance from the mucosal margin to the bottom of the probeable pocket in mm. A mean value will be calculated for each implant as well as for each subject. PPD changes in millimetres at the 10 year follow-up visit will be compared to values obtained at delivery of permanent restoration. Negative value denotes deeper pocket depth.
Time Frame: Time of permanent restoration and 10 years after permanent restoration
Population: Follow-up Extension (10 years) cohort. At visit 15 (10-year follow-up visit) 29 subjects remained in the short implants group, and 32 subjects remained in the long implants group. All subjects were included in the ITT population and were included in the analysis of PPD.
Measure: Mean (Standard Deviation); unit: Millimetre
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 29 | 32
Millimetre | -0.4 (1.2) | -0.7 (1.5)

8. Secondary Outcome: Change in Overall Oral Health Impact Profile (OHIP-49)
Description: OHIP-49 is describing the consequences of different oral diseases and conditions. It contains 49 items (questions) divided into 7 domains which are; functional limitation, pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. OHIP-49 attempts to measure both the frequency and severity of oral problems on functional and psychosocial well-being. Responses are based on a Likert response, with scale range; 0 = never, 1 = hardly ever, 2 = occasionally, 3 = fairly often, 4 = very often, for each of the 49 questions with a higher score being related to a worse outcome. To facilitate assessment of perceived severity of impacts, each statement has a weight derived using the Thurstone's paired comparison technique to reflect the relative importance of each statement. The overall OHIP-49 include all 49 questions with a total minimum score of 0 and a maximum total score of 196, with a higher score being related to a worse outcome.
Time Frame: At baseline (Visit 1 - screening and pre-surgical planning visit) and 5 years after permanent restoration
Population: Initial study (5 years) cohort. At visit 10 (5-year follow-up visit) 44 subjects remained in the short implants group, and 46 subjects remained in the long implants group. All subjects with available OHIP-values from baseline and 5 years after permanent restoration were included in the analysis of overall OHIP-49.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 33 | 35
score on a scale | -12 (26.3) | -16.9 (23.9)

9. Secondary Outcome: Change in Overall Oral Health Impact Profile (OHIP-49)
Description: as for outcome 8
Time Frame: At baseline (Visit 1 - screening and pre-surgical planning visit) and 10 years after permanent restoration
Population: Follow-up Extension (10 years) cohort. At visit 15 (10-year follow-up visit) 29 subjects remained in the short implants group, and 32 subjects remained in the long implants group. All subjects with available OHIP-values from baseline and 10 years after permanent restoration were included in the analysis of overall OHIP-49.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Short Implants | Long Implants in Combination With Bone Grafting
Number analyzed (Participants) | 15 | 16
score on scale | -2.2 (19.1) | -9.8 (16.3)

ADVERSE EVENTS:
Time Frame: From enrollment up to study termination, i.e. up to 5 years post permanent restoration for subjects not consenting to the study prolongation, and up to 10 years post permanent restoration for the 10-years extension cohort.
Groups:
- Short Implants - All Subjects, Including the 10-years Extension Cohort: ASTRA TECH Implant System, OsseoSpeed™ 4.0 S (length: 6 mm)
- Long Implants + Grafting - All Subjects, Including the 10-years Extension Cohort: ASTRA TECH Implants System, OsseoSpeed™ implants (lengths: 11, 13, 15 mm) in combination with grafing
Arm/Group | Short Implants - All Subjects, Including the 10-years Extension Cohort | Long Implants + Grafting - All Subjects, Including the 10-years Extension Cohort
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 6/50 | 7/51
Other Adverse Events (participants affected / at risk) | 23/50 | 27/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Implants - All Subjects, Including the 10-years Extension Cohort (N=50) | Long Implants + Grafting - All Subjects, Including the 10-years Extension Cohort (N=51)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Aorta stent (Cardiac disorders) | 0 (0) | 1 (1)
Knee replacement surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Car accident, back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain during dental surgery procedure (Cardiac disorders) | 0 (0) | 1 (1)
Benign medular tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blood cancer (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Fracture left shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hematoma upper leg (hospitalization) (Vascular disorders) | 0 (0) | 1 (1)
Heart valve replacement (Cardiac disorders) | 1 (1) | 0 (0)
Pancreas cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leg fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Implants - All Subjects, Including the 10-years Extension Cohort (N=50) | Long Implants + Grafting - All Subjects, Including the 10-years Extension Cohort (N=51)
Abutment related event (Product Issues) | 12 (17) | 10 (11)
Swollen after oral surgery (Investigations) | 3 (3) | 8 (8)
Crown related event (Product Issues) | 8 (11) | 9 (9)
Hypertension (Cardiac disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No